CLINICAL TRIAL: NCT03309501
Title: Study on Efficacy, Safety and Economy of Tong-Luo-Qu-Tong Plaster Treatment for Knee Osteoarthritis: Study Protocol for a Randomised, Double-blind, Parallel Positive Control, Multi-center Clinical Trial
Brief Title: Tong-Luo-Qu-Tong Plaster for KOA: a Randomised, Double-blind, Parallel Positive Control, Multi-center Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); Luoyang Osteopathy hospital of Henan (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); Liaoning University of Traditional Chinese Medicine (Other); The Second Hospital of Nanjing Medical University (Other); The Fourth Central Hospital of Tianjin (Unknown)
Responsible Party: Principal Investigator, Cui xuejun, associate professor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLQT Plaster
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis; Chronic Musculoskeletal Disease
Keywords: Knee osteoarthritis; Randomised Double-blind Controlled trial; Tong-Luo-Qu-Tong Plaster
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: positive control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tong-Luo-Qu-Tong Plaster group (Experimental): Intervention: Tong-Luo-Qu-Tong Plaster, daily 1 time, conventional treatment lasted for 14 days as two courses
  Interventions: Drug: Tong-Luo-Qu-Tong Plaster
- Qi-Zheng-Xiao-Tong Plaster group (Active Comparator): Intervention: Qi-Zheng-Xiao-Tong Plaster, daily 1 time, conventional treatment lasted for 14 days as two courses
  Interventions: Drug: Qi-Zheng-Xiao-Tong Plaster

INTERVENTIONS:
Drug: Tong-Luo-Qu-Tong Plaster — for 14 days as two period of treatment, daily 1 time.
  Arms: Tong-Luo-Qu-Tong Plaster group
Drug: Qi-Zheng-Xiao-Tong Plaster — for 14 days as two period of treatment, daily 1 time
  Arms: Qi-Zheng-Xiao-Tong Plaster group

SUMMARY:
Knee osteoarthritis(OA), also known as degenerative arthritis, have affected a lot of people. Patients with severe osteoarthritis frequently develop one or more of the typically following symptoms: joint pain, stiffness, activity with joint friction noise, limited mobility, such as difficulty walking and climbing. Now there are many western medicine treatments including symptom relief and joint cartilage protective agents for OA, but the results have not yet satisfied. TCM treatment of osteoarthritis has remarkable curative effect and unique advantage.Tong-Luo-Qu-Tong Plaster is a common method to treat osteoarthritis of the knee for thousands of years in China. It lacked a large sample randomised, double-blind, parallel positive controlled, multicenter clinical trial, and the clinical evidence of Tong-Luo-Qu-Tong Plaster for Knee Osteoarthritis need to be further completed.

DETAILED DESCRIPTION:
A randomised, double-blind, parallel positive controlled, multicenter clinical trial will be conducted to assess the effectiveness and safety of Tong-Luo-Qu-Tong Plaster on patients with knee osteoarthritis. A total of 2000 patients with knee osteoarthritis will be recruited and randomly allocated into experimental group(1500) or control group(500). Each patient will undergo a 2-week treatment with herbal patches for one session per day.The western Ontario and McMaster universities osteoarthritis index (WOMAC) as objective indicators of efficacy is the primary efficacy endpoint of the study.The secondary outcome measures are the changes in TCM syndrome quantitative score, Visual Analog Scale/Score (VAS) score of pain, and the effective time of pain relief of drug from the baseline to 1 week, 2 weeks' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have symptomatic knee osteoarthritis, diagnosis of KOA was based on criteria developed by the American College of Rheumatology(ACR) in 1986
* The differentiation standard of the arthralgia syndrome of traditional Chinese medicine(TCM): Referring to the Guidelines on the clinical research of Chinese medicine new drugs(2002)
* The visual analog scale score is no less than 30 mm.
* The patient is older than or equal to 40 years old
* All the patients signed informed consent form before study begins

Exclusion Criteria:

* Hormone therapy was used in the first month of screening
* Arthroscopy and intra-articular injection was performed on the knee joint which is going to be evalued during the first three months of screening.
* There is a history of trauma or surgery in the knee joint six months before screening or participants who a history of lessmore than three trauma or surgical procedures in the knees
* Participants who have knee arthroplasty, lumbar spinal stenosis, ankylosing spondylitis, rheumatic arthritis, rheumatoid factor positive(>40), eallergic constitution and mental disorder will be excluded from the trial
* Patients has severe diseases and complications such as severe diabetes, serious liver and kidney disease, malignant tumors, infectious diseases or complications affecting the knee joints
* Pregnant,lactating women
* Subjects are participating in or have participated in other clinical trials in the first three months.
* Subjects cannot stop using the drugs immediately with a long-term use of other related drugs.
* Combined with severe primary diseases such as hepatic renal functionand hematopoietic system, such as liver function (ALT≧1.5×ULN), and kidney function(AST≧1.5×ULN)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
WOMAC scores | from baseline to 2 weeks
  Western Ontario and McMaster universities osteoarthritis index, ranges 0-96. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
TCM syndrome quantitative scores | from baseline to 2 weeks
  Referring to the Guidelines on the clinical research of Chinese medicine new drugs(2002), the TCM syndrome quantitative score ranges 0-21.Higher values represent a worse outcome.
Visual analogue pain scale | from baseline to 2 weeks
  Visual Analog Scale /Score ranges 0-10.Higher values represent a worse outcome.
On effective time of pain relief of drug | In 2 weeks
  The effective time of pain relief was the time of 10mm was reduced for the first time according to the daily VAS score of the patient's diary.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Doctor, Principal Investigator — Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu BP, Yao M, Tian ZR, Zhou LY, Yang L, Li ZJ, Zhu S, Wang XT, Lan JH, Wang YJ, Cui XJ. Study on efficacy and safety of Tong-luo Qu-tong plaster treatment for knee osteoarthritis: study protocol for a randomized, double-blind, parallel positive controlled, multi-center clinical trial. Trials. 2019 Jun 24;20(1):377. doi: 10.1186/s13063-019-3481-6. PMID 31234919